CLINICAL TRIAL: NCT05538780
Title: Thoracic Fluid Content Using Electrical Cardiometry Versus Lung Ultrasound in the Diagnosis of Transient Tachypnea of Newborn
Brief Title: Diagnosis of Transient Tachypnea of Newborn
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ashraf Mohamed Ibrahim, clinical professor, Tanta University
Other Study IDs: 34987/10/21
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Transient Tachypnea of the Newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Transient tachypnea of the newborn (TTN) is the most common cause of respiratory distress in fullterm newborn. TTN is a diagnosis of exclusion, It is primarily diagnosed based on medical history and typical clinical presentation. Lung ultrasonography is an accurate, non invasive and reliable tool for diagnosing TTN. Cardiometry is presently the only tool to evaluate thoracic fluid content continuously and noninvasively at the bedside.

ELIGIBILITY:
Inclusion Criteria:

* fifty newborns with gestational age ≥ 34 weeks (calculated from the first day of last menstrual period and using New Ballard score) diagnosed with TTN

Exclusion Criteria:

1. Gestational age less than 34 weeks.
2. Major congenital abnormalities.
3. Congenital heart diseases.
4. Neonatal sepsis.
5. Neonatal pneumonia.
6. Other causes of respiratory distress (RD)

Ages: 0 Days to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 50 neonates diagnosed with Transient Tachypnea of Newborn admitted at Neonatal Intensive Care Unit, Tanta University Hospitals
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
change of thoracic fluid content | at enrollment and after 72 hours of birth
  measured by electrical cardiometry ( ICON®; Osypka Medical, Berlin, Germany)
change of ultrasound data: double-lung point, interstitial lung syndrome, and fuzziness of the pleural lines (A-lines) and pleural effusion. | at enrollment and after 72 hours of birth
  using Siemens Acuson X300 ultrasound machine ( Siemens Health Care GmbH, Erlangen, Germany )

CONTACTS AND LOCATIONS:
Overall Officials: ashraf abuhamama, Study Director — Tanta university faculty of medicine
Locations (1):
- Tanta University, faculty of medicine, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hammad Y, Hasanin A, Elsakka A, Refaie A, Abdelfattah D, Rahman SA, Zayed M, Hassabelnaby Y, Mukhtar A, Omran A. Thoracic fluid content: a novel parameter for detection of pulmonary edema in parturients with preeclampsia. J Clin Monit Comput. 2019 Jun;33(3):413-418. doi: 10.1007/s10877-018-0176-6. Epub 2018 Jun 23. PMID 29936563
- [Background] Paviotti G, De Cunto A, Moressa V, Bettiol C, Demarini S. Thoracic fluid content by electric bioimpedance correlates with respiratory distress in newborns. J Perinatol. 2017 Sep;37(9):1024-1027. doi: 10.1038/jp.2017.100. Epub 2017 Jul 27. PMID 28749485
- [Background] Ibrahim M, Omran A, AbdAllah NB, Ibrahim M, El-Sharkawy S. Lung ultrasound in early diagnosis of neonatal transient tachypnea and its differentiation from other causes of neonatal respiratory distress. J Neonatal Perinatal Med. 2018;11(3):281-287. doi: 10.3233/NPM-181796. PMID 30040751